CLINICAL TRIAL: NCT01716130
Title: Acceptability of Fluzone Intradermal Vaccine to Patients and Vaccine Administrators
Status: Completed | Type: Observational
Sponsor: Touro University, California (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, James E. Foy, D.O., Professor of Pediatrics, Touro University College of Osteopathic Medicine, Touro University, California
Other Study IDs: M0611
Record Dates: First submitted 2012-10-24; First posted 2012-10-29 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Patient Response to Fluzone ID Vaccine
Keywords: Fluzone Intradermal vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- IM vaccine in the past 3 years: Those subjects that received the Fluzone ID influenza vaccine, and reported having received the IM influenza vaccine in the past three years.
- no IM vaccine in the past 3 years: Patients that received the Fluzone ID vaccine and reported not receiving the IM influenza vaccine in the past 3 years.
- vaccine administrators: Those experienced vaccine administrators that administered the Fluzone ID vaccine, and were then surveyed concerning safety and overall satisfaction with the ID vaccine in comparison to the IM vaccine.

SUMMARY:
To assess the acceptance of the Fluzone Intradermal (ID)vaccine in adults and vaccine administrators in the United States. Patients completed 2 surveys, one immediately post-vaccination and one seven days later, that documented demographics and assessed their injection pain, injection anxiety, speed of injection, overall satisfaction, and preference for next year's vaccine. Vaccine administrators completed one survey assessing ease of vaccine preparation and administration, time required to administer, and safety/risk of needle stick injury for patient and administrator.

DETAILED DESCRIPTION:
Patients were divided into two groups: 1) those that reported receiving the intramuscular (IM) influenza vaccine in the past 3 years; and 2) those that reported not receiving the IM influenza vaccine in the past 3 years. The survey responses were compared between the two groups. In addition, the subjects that reported receiving the IM vaccine in the past 3 years were asked to compare their experience with the IM vaccine versus the ID vaccine.

ELIGIBILITY:
Inclusion Criteria:Age 18 -64 years of age Desire to receive the Fluzone Intradermal vaccine to protect against influenza. -

Exclusion Criteria:Less than 18 years of age, or 65 years of age and older. Desire to receive the Fluzone Intramuscular vaccine to protect against influenza.

problems of the immune system, current illness, severe allergy to eggs, severe (life threatening) allergies, history of having Guillain-Barre Syndrome (a severe paralytic illness) or having received a flu vaccine in the past three months.

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Overall patient satisfaction with intradermal vaccine | 7 days
  Overall patient satisfaction was assessed immediately post-vaccination and seven days later by patient survey.

SECONDARY OUTCOMES:
Overall satisfaction with the Fluzone ID vaccine by vaccine administrators | seven days
  Vaccine administrators (#8)completed a survey rating the ID vaccine in comparison to the IM vaccine in terms of ease of vaccine preparation, time required to administer the vaccine, and safety/needle stick risk for patients and administrators.

OTHER OUTCOMES:
Overall satisfaction with the Fluzone ID vaccine in two cohort groups | 7 days
  Using a survey tool, patients receiving the Fluzone ID vaccine were separated into 2 groups: 1) those that reported receiving the IM influenza vaccine in the past 3 years; and 2) those that reported not receiving the IM influenza vaccine in the past 3 years. All subject's satisfaction was assessed by survey immediately post-vaccination and 7 days later. Survey responses were compared between the 2 groups. The group that reported receiving the IM influenza vaccine in the past 3 years was asked to compare their experience with the ID vaccine in comparison to the IM vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: James E Foy, D.O., Principal Investigator — Touro University, California
Locations (1):
- Touro University California, Vallejo, California, United States

REFERENCES:
- See also: Touro University California Web Site — http://www.tu.edu